CLINICAL TRIAL: NCT06842225
Title: Interactive Roles of Cardiorespiratory Fitness and Adiposity on Recovery of Impaired Glucose and Vascular Control After Physical Inactivity
Brief Title: Interactive Roles of Cardiorespiratory Fitness and Adiposity on Glucose and Vascular Control After Physical Inactivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miami University (Other)
Responsible Party: Principal Investigator, Kevin Ballard, Principal Investigator, Miami University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 02290-1R15HL177798-01
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Disorders; Physical Inactivity; Vascular Disease Risk
Keywords: physical activity; glucose control; vascular function
MeSH Terms: conditions — Metabolic Diseases; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: We will recruit, screen, and enroll eligible participants (18-40y) across the following four groups: high CRF/low adiposity; high CRF/high adiposity; low CRF/low adiposity; low CRF/high adiposity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced physical activity (Experimental): We will recruit, screen, and enroll eligible participants (18-40y) across the following four groups: high CRF/low adiposity, high CRF/high adiposity; low CRF/low adiposity; low CRF/high adiposity. Each participant will undergo a three-week study. For the first week, participants will be instructed to maintain their normal level of physical activity. For the second week, participants' schedules will be examined, and strategies designed to reduce steps (by at least 2000 steps) and physical activity. To assist in reducing walking and increased sitting, participants will be given seated electric scooters to use whenever they normally walk. The scooters will be returned on the third week, and participants will be instructed to resume their normal physical activity. During the entire three weeks, participants will wear a continuous glucose monitor and a physical activity monitor.
  Interventions: Other: reduced physical activity

INTERVENTIONS:
Other: reduced physical activity — Each participant will undergo a three-week study. For the first week (day -7 to day 0), participants will be instructed to maintain their normal level of physical activity. For the second week (day 0 to day 7), the reduced physical activity (RPA) week, participants' schedules will be examined, and strategies designed to reduce steps (by at least 2000 steps) and physical activity (by taking elevators and short-cuts, etc.) by increasing sitting time >10%. To assist in reducing walking and increased sitting, participants will be given seated electric scooters to use whenever they normally walk. The scooters will be returned on the third week (day 7 to day 14), and participants will be instructed to resume their normal physical activity. During the entire three weeks, participants will wear a continuous glucose monitor (CGM) and a physical activity monitor (ActivPal).

SUMMARY:
The far-reaching negative health effects of the reduced physical activity (RPA) epidemic are often overlooked by the general population and health professionals. Short-term RPA induces cardiometabolic dysfunction, including impaired glucose control and vascular function, that may precede disease development. The impact of existing health status on RPA-induced cardiometabolic dysfunction and recovery of impaired glucose control following RPA is unexplored. Thus, the investigators' objectives are 1) to investigate the effect of existing health status (cardiorespiratory fitness and adiposity) on the recovery of impaired glucose control following a period of RPA and 2) to determine the role of vascular function as a mechanism of impaired glucose control. The investigators' final objective is to 3) expose undergraduate students to meritorious biomedical clinical research methods. The investigators have piloted the clinical research methods and analysis with undergraduate researcher associates and are well-prepared to complete this proposal. Preliminary data show that low cardiorespiratory fitness and/or high adiposity impair the recovery of glucose control following short-term RPA. Thus, the investigators aim to examine the interactive role of health status (cardiorespiratory fitness and adiposity) on the ability to recover impaired glucose control following short-term RPA. The investigators also seek to examine changes in vascular function as a mechanism of recovery of impaired glucose control following a return to normal PA. The investigators will recruit men and women with divergent health status (cardiorespiratory fitness and adiposity) to examine glucose control and vascular function during 7-d of normal PA, 7-d of RPA, and 7-d of resumption of normal RA. Continuous glucose monitoring and oral glucose tolerance tests will be performed to assess glucose control. Increases in vascular shear stress induced by passive leg movement and central arterial stiffness will be measured to assess vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 40 years of age.
* Ability to safely ride an electric scooter (e-scooter) for at least 10 minutes.
* Active (>7000 steps per day, walking > 1 mile a day outside)
* Stable body weight for at least 1 year
* aerobic fitness level, CRF is < 9 and >14 METS
* Visceral adipose tissue <130 cm2 or ≥130 cm2 for men and <100 cm2 or ≥100 cm for women

Exclusion Criteria:

* Any injury preventing them from exercising regularly at the time of the screening.
* Implantable defibrillator or pacemaker
* Active cancer
* Alcohol or drug abuse
* Use of an assistive walking device
* Presence of significant signs/symptoms of cardiovascular, metabolic, or pulmonary disease (determined from the American College of Sports Medicine (ACSM) Health History Questionnaire)
* Daily vitamin consumption of > 500mg per day during the study
* Acetaminophen or aspirin use during the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Daily Physical Activity | 3 weeks
  Accelerometers will be use to measure changes in daily physical activity during the three week study duration. Accelerometer data to be reported includes: daily number of steps, daily sitting time, daily stepping time, total sedentary time, and activity score.
Oral Glucose Tolerance Test (OGTT) | Days 0, 7, and 14
  On the morning of each OGTT, participants will arrive in the lab following an 8-10 h fast. An indwelling intravenous catheter will be placed into a forearm vein. Baseline (0 min) blood samples will be collected into heparinized evacuated tubes following 15 min of seated rest. Participants will consume a volume of glucose tolerance beverage containing 1 gram of glucose/kg of lean body mass to control for expected differences in body and fat mass between individuals. Participants will remain rested in the reclined position for the duration of the OGTT. Blood samples will be collected at 30, 60, 90, and 120 min post drink. Heparinized blood samples will be utilized to assess blood glucose using the Contour Next blood glucose monitoring system.
Continuous Glucose Monitoring | 3 weeks
  Participants will wear CGM sensors for the duration of the study, with the first sensor being placed on day -7 and a second sensor replacing it on day 0. Data will be exported and quality-checked data will be imported into the IGlu Application in R Studio and analyzed using the following parameters: Night hours set from 10 PM to 7 AM; Time above (high) set to 140 mg/dL; Time above (low) set to 120 mg/dL; Time in range set to 70-120 mg/dL; Time below (high) set to 70 mg/dL; Time below (low) set to 54 mg/dL; Data reported using this software includes weekly and daily means, standard deviations (SD), coefficient of variations (CV), medians, time below range < 54 mg/dL (TBR <54), time below range < 70 mg/dL (TBR <70), time in range 70-120 mg/dL (TIR 70-120), time above range >120 mg/dL (TAR >120), time above range >140 mg/dL (TAR >140), mean amplitude of glycemic excursions (MAGE), and area under the curve (AUC).
Femoral Artery Blood Flow | Days 0, 7, and 14
  Passive leg movement (PLM)-induced reactive hyperemia will be measured to assess peripheral vascular function. Briefly, the PLM technique involves passive movement of the leg to elicit a reactive hyperemic response measured by high-frequency ultrasonographic imaging. Diameter and blood velocity in the common femoral artery will be measured following 15 minutes of seated rest using a 5 to 12MHz multi-frequency linear array transducer connected to a high-resolution ultrasound. Arterial diameter and velocity will be recorded continuously for 60 seconds at baseline and 60 seconds during PLM. Femoral artery blood flow and shear rate (estimate of shear stress) will be calculated from arterial diameter and blood velocity measurements.

SECONDARY OUTCOMES:
Fat Mass and Fat-Free Mass | Days 0, 7, and 14
  Fat mass (kg) and fat-free mass (kg) will be determined using bioelectrical impedance and dual x-ray absorptiometry.
Height | Days 0
  Height (cm) will be determined using a wall-mounted stadiometer.
Central Arterial Stiffness | Days 0, 7, and 14
  Carotid-femoral pulse wave velocity will be measured following 10 min of rest to assess central arterial stiffness.
Central Arterial Blood Pressure | Days 0, 7, and 14
  Pulse wave analysis will be measured following 10 min of rest to assess central arterial blood pressure.
Blood Lipids | Days 0, 7, and 14
  A blood sample will be collected during fasted conditions on Days 0, 7, and 14 for determination of blood lipids (total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and triglycerides).
Cardiorespiratory Fitness | Day 0
  On the screening day, participants will perform a Balke-graded exercise treadmill test to assess cardiorespiratory fitness. This test will be conducted on a treadmill and lasts between about 10 and 20 minutes. Heart rate, oxygen consumption, and rating of perceived exertion (RPE) will be monitored every minute during the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Phillips Hall, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

DOCUMENTS (1):
  • Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT06842225/ICF_000.pdf